CLINICAL TRIAL: NCT05011357
Title: Effect of Phenylephrine Infusion on Pulse Pressure Variability
Brief Title: Phenylephrine and Pulse Pressure Variability
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Texas Health Resources (Other)
Responsible Party: Principal Investigator, Noah Jouett, Resident Anesthesiologist, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STU-2021-0497
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Intraoperative Hypotension
Keywords: Phenylephrine; Pulse pressure variation
MeSH Terms: interventions — Phenylephrine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phenylephrine (Experimental): Phenylephrine infusion (0.3 mcg/kg/hr)
  Interventions: Drug: Phenylephrine
- Control (Placebo Comparator): Saline infusion
  Interventions: Drug: Saline Control

INTERVENTIONS:
Drug: Phenylephrine — Phenylephrine will be administered as an infusion
  Other Names: Phenylephrine infusion
  Arms: Phenylephrine
Drug: Saline Control — Saline infusion
  Other Names: Saline
  Arms: Control

SUMMARY:
The purpose of this research study is to determine how vasopressors affect a measure of how intravenous fluid is administered in people undergoing surgery who have low blood pressure called Pulse Pressure Variability (PPV). This study will recruit human subjects to undergo simulated hypovolemia called Lower Body Negative Pressure (LBNP) and will receive phenylephrine and placebo, while PPV will be measured in both conditions. This research will help anesthesiologists learn more about how to use PPV in patients undergoing surgery and who need vasopressors.

DETAILED DESCRIPTION:
Perioperative fluid administration is a very important issue in modern anesthesia practice. Overzealous intraoperative administration of fluids can lead to cardiac overload thus potentially causing significant morbidity. It has been demonstrated that over 50% of perioperative complications are tied to intraoperative fluid administration and that changing intraoperative fluid management alone has significant positive benefit. Pulse pressure variation (PPV), which quantifies the respiratory variation in beat-to-beat arterial blood pressure, is viewed as a reliable method to assess volume status. Increasing PPV indicates hypovolemia, and a decreasing PPV indicates progression towards euvolemia. However, there are many commonly encountered intraoperative conditions that may make these interpretations of PPV problematic. For example it is commonly accepted in the perioperative community that PPV is interpretable in patients without vasopressor infusion since there is little consensus to the effects of vasopressor therapy on PPV. Hence the proposed study seeks to characterize the PPV response during simulated hypovolemia with and without infusion of phenylephrine, which acts on alpha-1 receptors to increase systemic vascular resistance, and hence blood pressure.

In a patient under general anesthesia, a PPV cut-off of 13% indicates a positive response to fluid administration. However, this cut-off was based on studies that used a wide variety of vasopressor agents with different mechanisms. Furthermore, it is unclear how effective the current threshold is at predicting fluid responsiveness when vasopressors are added during the same operation (i.e. a PPV of 13% without vasopressors likely represents different physiologic conditions compared to a PPV of 13% with vasopressors in the same operation). Hence, understanding how vasopressors such as phenylephrine change PPV and the PPV threshold is very important and represents an important knowledge gap in the practice of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years of age
* Non-obese (Body Mass Index less than 30 kg/m2)
* Baseline systolic blood pressure between 80-140 mmHg
* Baseline diastolic blood pressure <90 mmHg

Exclusion Criteria:

* Participants who have cardiac, vascular, respiratory, neurological and/or metabolic illness
* Current or previous use of anti-hypertensive medications
* Any known history of renal or hepatic insufficiency/disease
* Pregnancy (verified by negative urine test on the experimental days) or breast-feeding
* Current smokers, as well as individuals who regularly smoked within the past 3 years
* Sulfite allergy, as this is a contraindication to intravenous phenylephrine
* Serious mental illness including claustrophobia
* History of use of recreational drugs including cocaine or amphetamines
* Peripheral vascular disease
* Subject on anticoagulant treatment
* Subjects with a baseline systolic blood pressure <80 mmHg

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Pulse Pressure Variability | Thirty minutes following phenylephrine infusion
  Quantifying respiratory variation in beat-to-beat arterial blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Noah Jouett, DO/PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Texas Health Resources, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No